CLINICAL TRIAL: NCT02253381
Title: Effect of Position During Spinal Anesthesia on Hemodynamic Change in Pregnant Women Undergoing Cesarean Section: Randomized Trial
Brief Title: Effect of Position During Spinal Anesthesia on Hemodynamic Change in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Panthila Rujirojindakul, Dr, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC: 57-195-08-1
Record Dates: First submitted 2014-09-27; First posted 2014-10-01 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hypotension
Keywords: lateral decubitus position; hypotension; cesarean section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right lateral decubitus position (Active Comparator): Right lateral decubitus position during spinal anesthesia
  Interventions: Procedure: Right
- Left lateral decubitus position (Active Comparator): Left lateral decubitus position during spinal anesthesia
  Interventions: Procedure: Left

INTERVENTIONS:
Procedure: Right — Right lateral decubitus position during spinal anesthesia
  Arms: Right lateral decubitus position
Procedure: Left — Left lateral decubitus position during spinal anesthesia
  Arms: Left lateral decubitus position

SUMMARY:
Hypotension is the most common complications after spinal anesthesia especially in pregnant patients who undergoing cesarean section. Position during spinal anesthesia may be altering the hemodynamic. For right lateral decubitus, the enlarged uterus compresses inferior vena cava that may decrease venous return and cardiac output. This leads to hypotension.The hypothesis is the right lateral position during spinal anesthesia in pregnant women will be had hemodynamic changing more than the left lateral position. This objective is to compare hemodynamic change between left and right lateral position during spinal anesthesia in pregnant women undergoing cesarean section.

DETAILED DESCRIPTION:
Study design: A randomized controlled trial

Study setting:

The study will be conducted in the operating rooms at Songklanagarind Hospital, Faculty of Medicine, Prince of Songkla University, Songkhla, Thailand

Study period:

The total duration of participation in the randomized study is up to the operative day.

Study population:

Pregnant patients undergoing cesarean section receiving spinal anesthesia with 0.5% bupivacaine and 0.2 mg morphine total volume 2.2 ml.

Study sample:

Inclusion criteria

1. Signed informed consent
2. Pregnancy
3. Spinal anesthesia with 0.5% bupivacaine and 0.2 mg morphine total volume 2.2 ml
4. Elective and emergency surgery

Exclusion criteria

1. Contraindication for spinal anesthesia
2. Complicated pregnancy such as maternal heart disease, eclampsia, severe fetal distress, abruption placenta, twin pregnancy, and placenta previa totalis
3. Maternal height < 150 cm.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Term pregnancy
* Spinal anesthesia with 0.5% bupivacaine and 0.2 mg morphine total volume 2.2 ml

Exclusion Criteria:

* Contraindication for spinal anesthesia
* Height < 150 cm.
* Complicated pregnancy e.g. heart disease, preclampsia, eclampsia, diabetes millitus, twin, abrupt placenta, placenta pre via, and fetal distress
* Failed spinal anesthesia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hypotension | after bupivacaine injection until 15 minutes after spinal anesthesia
  Systolic blood pressure lower than 90 mmHg or decrease more than 20% of baseline

SECONDARY OUTCOMES:
Ephedrine consumption | intraoperative
  Total amount of ephedrine receiving
Apgar score at first minute and fifth minute | Child delivery at first minute and fifth minute

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanish, MD, Study Chair — Ethical Committee
Locations (1):
- Department of anesthesiology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand